CLINICAL TRIAL: NCT02712125
Title: Nitric Oxide Donors for Treatment of Isolated Oligohydramnios: A Pilot Study
Brief Title: Nitric Oxide Donors for Treatment of Isolated Oligohydramnios
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Benha University (Other)
Responsible Party: Principal Investigator, Ahmed Walid Anwar Murad, Assistant Professor, Department of Obstetrics and Gynecology, Faculty of Medicine, Benha University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Benha-023
Record Dates: First submitted 2016-03-02; First posted 2016-03-18 (Estimated); Last update posted 2016-03-18 (Estimated); Status verified 2016-03

CONDITIONS: Isolated (Idiopathic) Oligohydramnios
MeSH Terms: conditions — Oligohydramnios | interventions — isosorbide-5-mononitrate; Tablets

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- isosorbide mononitrate (Active Comparator): Received 20 mg isosorbid mononitrate (IMN) (Effox, Mina Pharma Co, Egypt; under license of Schwartz Pharma, Germany) vaginally once daily until delivery
  Interventions: Drug: isosorbide mononitrate
- Control (Placebo Comparator): Received placebo vaginal tablets once daily until delivery
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: isosorbide mononitrate — 20 mg isosorbide mononitrate (IMN) tablet applied vaginally once daily until delivery .
  Other Names: Effox 20 mg tablet
  Arms: isosorbide mononitrate
Drug: Placebo — placebo vaginal tablets once daily until delivery
  Arms: Control

SUMMARY:
Objective: To assess the influence of maternal isosorbide mononitrate (IMN) vaginal supplementation in improving liquor volume in women with isolated oligohydramnios.

Study Design: Prospective randomized interventional study. Materials and Methods: 100 women with singleton pregnancy about 28-36 weeks, with isolated oligohydramnios [amniotic fluid index (AFI) < 5] were enrolled in the study. Before the proposed intervention, the antenatal risk factors were studied. Patients received 20 mg isosorbide mononitrate (IMN) vaginally. Patient were followed after 24 hours then weekly. The treatment was continued till the liquor improved significantly or until delivery. Outcome measures; mean increase in liquor, intervention delivery interval, and neonatal outcome were studied.

DETAILED DESCRIPTION:
This prospective randomized interventional study was done in Obstetrics and Gynecology Department , Benha University Hospital, Alkalubia, Egypt from August 2013 to August 2015.

The study protocol was approved by the Local Ethics Committee and written informed consents were taken from patients entering the study. The study included 100 women aged 18-35 years with singleton pregnancy about 28-36 weeks gestation, with diagnosed isolated oligohydramnios (AFI less than 5 cm).

Initially, all the participants were subjected to through routine antenatal history taking and examination and by routine ultrasound scan using (Voluson, 730 Pro V, GE Medical System), AFI was assessed. All participants were instructed to take regularly the daily water requirement, especially in the two days before starting the study and throughout the study. Participants were randomly scheduled into two equal groups by computer-generated blocks into a control group received placebo vaginal tablets and a study group received 20 mg isosorbide mononitrate (IMN) vaginally once daily until delivery (Effox, Mina Pharma Co, Egypt; under license of Schwartz Pharma, Germany). Treatment allocation was concealed by using sequentially numbered opaque sealed envelopes, opened sequentially by a third person (study nurse). Amniotic fluid index was rechecked after two days and followed up weekly till delivery by one person to avoid interobserver variability. Drug treatment continues until the volume of the fluid reach the normal value or until delivery. Antenatal vitamins were continued.

Primary outcome measure was the change in AFI.

Secondary outcome measures were the side effect of isosorbide mononitrate if any, indications and mode of delivery, and neonatal outcomes as regard birth weight, still birth or neonatal death, Apgar score and the need for neonatal admission.

ELIGIBILITY:
Inclusion Criteria:

* Singleton pregnancy
* 28-36 weeks gestation,
* Diagnosed isolated oligohydramnios (AFI less than 5 cm).

Exclusion Criteria:

* Multiple pregnancy;
* Fetal chromosomal or congenital abnormalities;
* Signs of fetal distress;
* Preterm rupture of membranes;
* Intrauterine infection;
* Receiving treatment for oligohydramnios ;
* History of maternal heart disease;
* Vasodilator use; sensitivity to NO donors ;
* Pre-existing chronic medical problems.

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2013-08; Primary Completion 2015-06 (Actual); Study Completion 2015-08 (Actual)

PRIMARY OUTCOMES:
The change in amniotic fluid index (AFI)in centimeters. | Through study completion, up to 40 weeks of gestations
  Technique of AFI measurement
  * Uterus is divided into four imaginary quadrants with linea nigra and umbilicus acting as the vertical and the horizontal axis respectively
  * The deepest pocket devoid of umbilical cord and fetal parts is measured in the vertical dimension
  * Measurement of the four pockets is in centimeters
  * Sum of all the four quadrant measurements is AFI
  * Normal AFI values range from 5 to 25 cm

SECONDARY OUTCOMES:
Number of participants with isosorbide mononitrate -related adverse events as assessed by CTCAE v4.0. | Through study completion, up to 40 weeks of gestations
Number of participants with each indication of delivery | Through study completion, up to 40 weeks of gestations
Number of participants with adverse neonatal outcomes | At time of delivery.
Number of participants delivered by Cesarean sections or vaginally | Through study completion, up to 40 weeks of gestations

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed Walid Anwar Murad, Principal Investigator — Department of Obstetrics and Gynecology, Faculty of Medicine, Banha University,